CLINICAL TRIAL: NCT06688786
Title: A Pospective, Single-arm, Multicenter Clinical Trial Evaluating Preoperative Neoadjuvant mFOLFOX6 Chemotherapy in Combination With PD1 Monoclonal Antibody in MSS/pMMR Locally Advanced Rectal Cancer (FIRM Study)
Brief Title: A Pospective, Single-arm, Multicenter Clinical Trial Evaluating Preoperative Neoadjuvant mFOLFOX6 Chemotherapy in Combination With PD1 Monoclonal Antibody in MSS/pMMR Locally Advanced Rectal Cancer
Acronym: FIRM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Tingyu Wu, Principal Investigator, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XHEC-C-2024-179-2
Record Dates: First submitted 2024-11-08; First posted 2024-11-14 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced Rectal Cancer (LARC)
Keywords: rectcal cancer; microsatellite stable; FOLFOX; neoadjuvant chemotherapy; PD-1 antibodies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combinational treatment group (Experimental): neoadjuvant mFOLFOX6 chemotherapy combined with PD-1 inhibitor therapy
  Interventions: Drug: neoadjuvant mFOLFOX6 chemotherapy combined with PD-1 inhibitor therapy

INTERVENTIONS:
Drug: neoadjuvant mFOLFOX6 chemotherapy combined with PD-1 inhibitor therapy — Preoperative treatment with 4-6 cycles of mFOLFOX6 regimen combined with serplulimab

SUMMARY:
Preoperative neoadjuvant chemoradiotherapy can induce tumor regression and reduce the risk of postoperative recurrence, serving as the standard treatment for locally advanced rectal cancer. However, neoadjuvant radiotherapy may increase the risk of postoperative complications, proctitis, enteritis, and reduced anal function. Exploring radiation-free approaches to prevent the effects of radiotherapy toxicity on postoperative complications and quality of life is now a significant research focus. Neoadjuvant chemotherapy represents a promising approach in the neoadjuvant treatment of rectal cancer. Neoadjuvant chemotherapy avoids the impact of radiotherapy on organ function, reduces the incidence of postoperative anastomotic leakage, and is beneficial for long-term anal function preservation. However, its low tumor regression rate limits its application in the neoadjuvant treatment of rectal cancer. For patients with locally advanced rectal cancer, there is an urgent need for a new neoadjuvant treatment strategy that can both significantly improve tumor regression rates and reduce the risk of postoperative anastomotic leakage, and protect long-term anal function. PD-1 inhibitors are highly effective in treating microsatellite instability-high (MSI-H) colorectal cancer patients, but show poor efficacy in the 95% of patients with microsatellite stable (MSS) tumors. The challenge now is to find combination therapies that can convert tumors into an "immune-activated tumor," thereby enhancing the effectiveness of immunotherapy in MSS patients. Oxaliplatin and 5-fluorouracil have roles in releasing tumor antigen epitopes, activating CD8+ cells, and reshaping the immune microenvironment. Multiple clinical studies and animal experiments have shown that combining PD-1 antibodies with FOLFOX generates a synergistic effect, showing strong antitumor activity. This study evaluates the efficacy, safety, and impact on postoperative anal function of preoperative neoadjuvant treatment with FOLFOX chemotherapy combined with PD-1 inhibitors in patients with MSS-type advanced rectal cancer. The radiotherapy-free approach aims to avoid radiotherapy-related toxicity, offering significant potential to enhance the efficacy of neoadjuvant chemotherapy, improve long-term survival, and protect anal function.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced (cT3-4NxM0 or cTxN+M0) rectal cancer with the lower tumor margin within 15 cm of the anal verge
2. Histopathology confirmed adenocarcinoma with an pMMR/MSS genetic profile.
3. Absence of bowel obstruction, or bowel obstruction relieved by proximal colostomy.
4. Age: 18-75
5. ECOG: 0-1
6. No prior chemotherapy, radiotherapy, targeted therapy, or immunotherapy received.
7. Female participants must be non-lactating, with a negative pregnancy test result.

Exclusion Criteria:

1. Patients with distant metastasis
2. History of receiving chemotherapy, radiotherapy, targeted therapy, or immunotherapy.
3. Active autoimmune disease requiring systemic treatment within the 2 years prior to enrollment.
4. History of other malignancies within the past 5 years, excluding cured cervical carcinoma in situ or basal cell carcinoma of the skin.
5. History of HIV infection, or active chronic hepatitis B or C with high viral DNA copy numbers.
6. Patients with active tuberculosis currently receiving anti-tuberculosis treatment or treated with anti-tuberculosis therapy within the past year prior to screening.
7. Known or suspected allergy to the study drug or any study-related medications administered.
8. Presence of severe cardiovascular or cerebrovascular disease.
9. Within 14 days prior to the first dose, presence of a severe active or uncontrolled infection requiring systemic therapy, or unexplained fever >38.5°C.
10. Receiving systemic corticosteroid treatment or other immunosuppressive agents within 14 days prior to the first dose, or immunostimulants within 4 weeks.
11. History of confirmed neurological or psychiatric disorders, including epilepsy or dementia.
12. The participant may be unable to complete the study due to other reasons, or the investigator considers them unsuitable for inclusion.
13. Refusal to sign the informed consent form.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response | Day 7 after surgery
Major Pathological Response | Day 7 after surgery

SECONDARY OUTCOMES:
Tumor regression grade | Day 7 after surgery
Radiologic Response | Preoperative evaluation
Neoadjuvant rectal score | Day 7 after surgery
  The Neoadjuvant rectal score ranges from 0 to 100, with higher scores indicating poorer response to neoadjuvant therapy.
Postoperative complication | Within 2 weeks post-surgery
Disease free survival | Three years after surgery
Relapse free survival | Three years after surgery
Wexner fecal incontinence scale | evaluated every 3 months for 3 years after surgery
  Utilized to evaluate anal function, with higher scores indicating poorer anal function.
overall survival | Three years after surgery
Adverse events | Prior to surgery, adverse events are evaluated the day before each chemotherapy cycle. After surgery, adverse events are evaluated at months 3, 6, 9, and 12.

CONTACTS AND LOCATIONS:
Locations (1):
- Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
In this study personal information and data such as patient history, physical examination results, surgical records, and study questionnaire data will be collected. These data will be used to evaluate the efficacy and safety of the therapeutic regimen and for academic publication. The researcher will treat the personal data of patients confidentially and anonymize the data and information in any public release of the results of the study.
Supporting Information: Study Protocol, SAP, CSR